CLINICAL TRIAL: NCT03666962
Title: Evaluating Medication Adherence to Novel Oral Anticoagulants With Anticoagulant Activity Monitoring in Patients With Atrial Fibrillation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cui Yimin (Other)
Responsible Party: Sponsor-Investigator, Cui Yimin, Director of pharmacy，M.D & Ph.D, Peking University First Hospital
Organization: Peking University First Hospital (Other)
Other Study IDs: 2018[136]
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Anticoagulants; Compliance, Medication
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Blood samples are divided into peak concentration and valley concentration. Peak concentration (Cmax) refers to the highest serum concentration after administration for at least one week in the study. Valley concentration (Cmin), the lowest concentration during administration, is usually obtained from the lowest concentration between the initial time of administration and the next time the drug is administered at a steady state (continuous medication for more than 1 weeks.).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case group: According to the scores of MGLS, compliance was divided into three groups: A score of 0 indicated high compliance; a score of 1 or 2 illustrated intermediate compliance; and a score of 3 or 4 indicated low compliance.
- control group: According to the scores of MGLS, compliance was divided into three groups: A score of 0 indicated high compliance; a score of 1 or 2 illustrated intermediate compliance; and a score of 3 or 4 indicated low compliance.

SUMMARY:
The novel oral anticoagulants such as rivaroxaban, apixaban and dabigatran, specifically target either thrombin or factor Xa/IIa. These new agents are included as an option for prevention of thromboembolic disease or recurrent stroke in patients with non-valvular atrial fibrillation in guidelines.

Although the benefits and risks of anticoagulation and antiplatelet therapy have been fully assessed, and reasonable anticoagulation and antiplatelet therapies have been formulated, the therapeutic effect still largely depends on the quality control during the treatment. Many patients discontinue anticoagulant therapy after discharge or after a period of treatment, and the risk of thrombosis increases. Because non-vitamin K antagonist oral anticoagulants (NOACs) does not need routine monitoring, patients tend to ignore the regular medication, thus affecting drug compliance. Because of the short half-life of NOACs, if patients do not take it regularly, not only can not achieve the effectiveness of anticoagulation, but also reduce the safety of medication. More and more researchers have realized that medication adherence plays a key role in medical management. In order to improve the efficacy and safety of NOACs and the compliance of patients with NOACs, the guidelines emphasize that supplementary measures can be taken, such as pharmacists participating in the network pharmacy database, attaching importance to the medication education of patients and their families, formulating a strict follow-up plan and professional outpatient follow-up.

DETAILED DESCRIPTION:
Patients with new oral anticoagulants will be included in the study. After the signing of the informed consent, blood samples were collected to detect the anti Xa factor activity after taking the drugs. Meanwhile, the medication compliance of the patients during the treatment was also collected.

Dedicated tests based on anti-Xa activity for rivaroxaban and apixaban and anti-IIa activity for dabigatran concentration was conducted. Blood samples are divided into peak concentration and valley concentration. Peak concentration (Cmax) refers to the highest serum concentration after administration for at least one week in the study. Valley concentration (Cmin), the lowest concentration during administration, is usually obtained from the lowest concentration between the initial time of administration and the next time the drug is administered at a steady state (continuous medication for more than 1 weeks.).

A compliance questionnaire was conducted to collect the compliance of the drug during treatment. The Morisky, Green, and Levine Adherence Scale (MGLS) was used to evaluate the medication adherence of non-vitamin K antagonist oral anticoagulants (NOACs) patients.

Based on the results of data analysis, the correlation between anti Xa/IIa activity test results and medication compliance was analyzed, making the anti Xa/IIa activity concentration a simple measure to predict the compliance of patients.

ELIGIBILITY:
Inclusion Criteria:

1. confirmed diagnosis of NOACs indications, such as thromboprophylaxis for non-valvular atrial fibrillation, prevention or treatment of deep vein thrombosis/pulmonary embolism, and thromboprophylaxis after knee/hip replacement.
2. Age >18 years old, unlimited for gender.
3. Written or phoned informed consent was obtained from all patients or their families.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who take NOACs at Peking University First Hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Pharmacodynamic indicators | at least 1 week after drug administration
  Blood samples are divided into peak concentration and valley concentration. Peak concentration (Cmax) refers to the highest serum concentration after administration for at least one week in the study. Valley concentration (Cmin), the lowest concentration during administration, is usually obtained from the lowest concentration between the initial time of administration and the next time the drug is administered at a steady state (continuous medication for more than 1 weeks.).
Medication adherence | at least 1 week after drug administration
  A compliance questionnaire was conducted to collect the compliance of the drug during treatment. According to the scores of MGLS, compliance was divided into three groups: A score of 0 indicated high compliance; a score of 1 or 2 illustrated intermediate compliance; and a score of 3 or 4 indicated low compliance.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - The Second Affiliated Hospital Of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The 7th People's hospital of the zhengzhou, Zhengzhou, Henan
  - Peking University First Hospital, Beijing
  - Beijing Hospital, Beijing
  - Fujian Medical University Union Hospital, Fuzhou
  - Fuzhou General Hospital of Nanjing Militray Command, Fuzhou
  - Anhui Provincial Hospital#The First Affiliated Hospital Of USTC#, Hefei

REFERENCES:
- [Derived] Liu Z, Xie Q, Xiang Q, Zhang H, Mu G, Zhao Z, Hu T, Wu T, Wang N, Zhang J, Qian Y, Zhou S, Wang Z, Jiang J, Zhang Y, Song H, Cui Y. Anti-FXa-IIa activity test in Asian and its potential role for drug adherence evaluation in patients with direct oral anticoagulants: a nationwide multi-center synchronization study. Cardiovasc Diagn Ther. 2020 Oct;10(5):1293-1302. doi: 10.21037/cdt-20-564. PMID 33224753